CLINICAL TRIAL: NCT00083876
Title: UARK 98-035, A Phase III Study of D.T. PACE Versus High Dose Melphalan and Autologous Transplant in Patients With Previously Treated Multiple Myeloma
Brief Title: D.T. PACE Versus High Dose Melphalan and Autologous Transplant in Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Edwina Mosby, CRA, University_of_Arkansas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-035
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; D.T. PACE; Melphalan; Transplant; Thalidomide; Dexamethasone; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Filgrastim; Interferon-alpha 2b; Sargramostim
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
This study has been designed to evaluate whether combination chemotherapy and "anti-angiogenesis" therapy with thalidomide is equal or superior to autologous transplantation for the treatment of multiple myeloma.

DETAILED DESCRIPTION:
All patients will receive two cycles, 4-6 weeks apart, of a combination of chemotherapy drugs (a regimen called D.T. PACE) and collection of peripheral blood stem cells. D.T. PACE consists of 6 chemotherapy drugs (Dexamethasone, Thalidomide, CisPlatin, Adriamycin, Cyclophoshamide, and Etoposide). Four to six weeks after the last cycle of D.T. PACE, each patient with no evidence of myeloma progression will be randomly assigned to receive 1) Autologous Transplant as described below or 2) Additional cycles of D.T. PACE. Since it is not known at this time which treatment is the best, patients will be placed by chance in one of the two groups. If tests show that myeloma is in remission at the time of randomization, 2 additional cycles of D.T. PACE will be given. If myeloma is not in remission, 2 additional cycles of D.T. PACE will be given, then the myeloma will be re-assessed. If the patients myeloma protein has decreased by 90% since baseline or better, 2 more cycles are given. If it has not decreased that much or has gotten worse, the patient will be offered autologous transplantation. Patients with no financial coverage for transplant, or those that have inadequate stem cell collections to support two transplants, will not be randomized and will proceed directly to treatment 2, continued D.T. PACE. If it is determined that the myeloma did not respond adequately to the first 2 cycles of D.T. PACE, then the patient will not be randomized and will proceed directly to autologous transplant.

Between 2 and 4 months after the first PBSC transplant, the patient will undergo a second course of high-dose Melphalan and PBSC transplant. In order for all patients to receive the maximum possible benefit, patients may "cross-over" to the other treatment arm if the myeloma does not go into complete remission or at any time myeloma progresses after randomization.

When the physician feels that the maximum benefit from chemotherapy has been received (best partial or complete remission) the last phase of the study will start, which is maintenance. Patients will be randomly assigned to receive either low dose (50 mg) or higher dose (200 mg) thalidomide with the dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have previously treated (> 1 cycle prior therapy), active multiple myeloma requiring treatment. Patients that have received >450 mg/m2 of prior Adriamycin therapy are eligible, however, Adriamycin will be deleted from the DT PACE regimen in these patients.
* Patients must have measurable disease defined as one of the following: serum monoclonal protein >/= 1.0 mg/dl, OR urine monoclonal protein >/= 1.0 grams/24 hour, OR >/= 20% bone marrow plasmacytosis.
* All necessary baseline studies for determining eligibility must be obtained within 35 days prior to registration.
* Patients must have a performance status of 0-2 based on SWOG criteria.Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* Patients must have a platelet count > or = 100,000/microliters. Patients with platelet count < 100,000/microliters may be enrolled if it is felt to be due to extensive marrow plasmacytosis. The study coordinator must be consulted and dose modifications may apply.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have received a prior autotransplant or allograft.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Patients with recent (< o= 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrythmias are ineligible. Ejection fraction by ECHO or MUGA should be within the institutional normal range and must be performed within 42 days prior to registration.
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease.Patients must have adequate pulmonary function studies > or = 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > or = 50% of predicted. Patients unable to complete pulmonary function tests due to myeloma related pain or fracture must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval and there must be no prior treatment with cytotoxic drugs that could potentially be assigned on this treatment protocol.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1998-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
1.1 To evaluate, in a randomized phase III clinical trial in previously treated multiple myeloma patients whether angio-chemotherapy with D.T. PACE may be equivalent or superior to tandem transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Barthel Barlogie, M.D., Ph.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675